CLINICAL TRIAL: NCT02213094
Title: Phase I Study of Nicotinamide for Early Onset Preeclampsia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: North Carolina Translational and Clinical Sciences Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 13-2203
Record Dates: First submitted 2014-08-07; First posted 2014-08-11 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-03

CONDITIONS: Pregnancy Induced Hypertension; Superimposed Preeclampsia; Hypertension
Keywords: preeclampsia; pregnancy-induced hypertension; nicotinamide
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Hypertension; Pre-Eclampsia | interventions — Niacinamide

STUDY DESIGN:
Intervention Model Description: Phase 1 dose escalation study
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Nicotinamide 500 mg (Experimental): Nicotinamide 500 mg by mouth each morning until delivery or 14 days, whichever occurs first.
  Interventions: Drug: Nicotinamide 500 mg
- Nicotinamide 1000 mg (Experimental): Nicotinamide 1000 mg by mouth each morning until delivery or 14 days, whichever occurs first.
  Interventions: Drug: Nicotinamide 1000 mg

INTERVENTIONS:
Drug: Nicotinamide 500 mg — Nicotinamide 500 mg taken by mouth each morning
  Other Names: Vitamin B3 amide
  Arms: Nicotinamide 500 mg
Drug: Nicotinamide 1000 mg — Nicotinamide 1000 mg taken by mouth each morning
  Other Names: Vitamin B3 amide
  Arms: Nicotinamide 1000 mg

SUMMARY:
This is a Phase I study of vitamin B3-amide (nicotinamide) dietary supplementation in pregnant women with early onset preeclampsia. The investigators will enroll 10 pregnant women at 24-32 weeks' gestation with the diagnosis of preeclampsia. If the woman is anticipated to remain undelivered for 48 hours after diagnosis she will receive vitamin B3-amide, 500 mg/day given in the morning (n=5) or 1000 mg given in the morning (n=5), continuing until delivery or for 14 days, whichever occurs first. Maternal blood will be collected at baseline and twice a day on days 1, 3, and 7 of nicotinamide administration to measure nicotinamide metabolites, The objectives of this Phase I study are to to test safety of nicotinamide.

ELIGIBILITY:
Inclusion Criteria:

1. Maternal age 18-45 years
2. Informed written consent
3. Preeclampsia or new onset hypertension between 24-32 completed weeks' gestation

   1. Hypertensive complications of pregnancy defined as new onset systolic BP > 140 mm Hg and/or diastolic BP > 90 mm Hg on two occasions 6 hours apart; OR > 300 mg proteinuria on 24 hour urine collection OR urine P/C ratio >0.3;
   2. Dating criteria based on menstrual dating confirmed by first or second trimester ultrasound OR second trimester ultrasound if menstrual dating unavailable;
   3. Deemed clinically stable by primary clinician and candidate for expectant management (delayed delivery);
4. Maternal liver function tests < 3x ULN
5. Maternal platelet count > 100,000 mm3
6. Fetal well-being established by estimated fetal weight > 5th %tile; normal amniotic fluid volume (MVP > 2 cm); normal Umbilical Artery Dopplers; AND reactive NST(non-stress test) or BPP (biophysical profile) > 6
7. Plan for expectant management until delivery
8. Delivery not anticipated within first 48 hours

Exclusion Criteria:

1. Preeclampsia < 24 or > 33 weeks' gestation;
2. Suspected fetal structural or chromosomal abnormality;
3. Pre-existing renal disease (creatinine > 1.5 mg/dL)
4. Pre-existing vascular disease (systemic lupus; cardiac disease;)
5. Plan for delivery within 48 hours
6. Any pre-existing medical condition that would increase risk for liver toxicity (e.g. hepatitis B or C; HIV)
7. Evidence of cerebral dysfunction (seizures; cerebral edema on CT/MRI; headache unresolved with oral analgesics)
8. Pulmonary edema
9. HELLP (hemolysis, elevated liver enzymes, low platelets syndrome)
10. Evidence of liver dysfunction (LFTs > 3x ULN)
11. Thrombocytopenia (platelets < 100,000 mm3)
12. Evidence of fetal compromise: EFW(estimated fetal weight) < 5th percentile; BPP < 6; absent or reverse diastolic UA blood flow; oligohydramnios (MVP < 2 cm)
13. Placental abruption defined as unexplained vaginal bleeding
14. Preterm labor defined as regular contractions and cervical change
15. Any condition deemed by the investigator to be a risk to mother or fetus in completion of the study
16. Any condition deemed by the investigator to require delivery within 48 hours

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2015-12-03 (Actual); Study Completion 2015-12-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim A Boggess, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Women's Hospital, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nicotinamide 500 mg | Nicotinamide 1000 mg
Started | 5 | 5
Completed | 4 (One subject stopped study agent early because of elevation in LFTs > 3x ULN) | 5
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nicotinamide 500 mg | Nicotinamide 1000 mg | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 5 | 10
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: Specific adverse events were Maternal liver toxicity, defined as > 3x ULN of ALT(Alanine amniotransferase) or AST (Aspartate amniotransferase), maternal report of side effects, and fetal adverse effects.
Time Frame: Within 48 hours of dosing
Measure: Number; unit: participants
Arm/Group | Nicotinamide 500 mg | Nicotinamide 1000 mg
Number analyzed (Participants) | 5 | 5
participants | 2 | 0

ADVERSE EVENTS:
Time Frame: During study agent administration (up to 14 days)
Arm/Group | Nicotinamide 500 mg | Nicotinamide 1000 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 2/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotinamide 500 mg (N=5) | Nicotinamide 1000 mg (N=5)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) — Subject #5 required dialysis following delivery of her infant. Her serum creatinine was normal at enrollment and throughout study agent administration. She developed renal failure following delivery, which required 2 dialysis treatments.
Elevated LFTs (Hepatobiliary disorders) | 1 (1) | 0 (0) — Subject #4 had elevated LFTs < 24 hours after first dose of study agent. This was believed to be due to the disease process and thus the primary clinical provider opted to proceed with infant delivery, therefore study agent was discontinued.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No